CLINICAL TRIAL: NCT02699723
Title: Oral Arsenic Trioxide and Itraconazole for the Treatment of Patients With Advanced Basal Cell Carcinoma
Brief Title: Arsenic Trioxide and Itraconazole in Treating Patients With Advanced Basal Cell Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Logistics
Sponsor: Jean Yuh Tang (Other)
Responsible Party: Sponsor-Investigator, Jean Yuh Tang, Associate Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-35488; NCI-2016-00180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKIN0033 (Other: Stanford Cancer Institute)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Skin Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Arsenic Trioxide; arsenous acid; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (arsenic trioxide, itraconazole) (Experimental): Patients receive arsenic trioxide PO and itraconazole PO daily for 50 days, followed by maintenance therapy consisting of 2 weeks off treatment and then 2 weeks on treatment for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Arsenic Trioxide; Drug: Itraconazole; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Arsenic Trioxide — Given PO
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid; Arsenous Acid Anhydride; Arsenous Oxide; Trisenox; White Arsenic
Drug: Itraconazole — Given PO
  Other Names: Lozanoc; Oriconazole; R 51,211; Sporanox
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well arsenic trioxide and itraconazole work in treating patients with basal cell cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Itraconazole may help treat fungal infections in patients with basal cell cancer. Giving arsenic trioxide with itraconazole may work better in treating basal cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response of arsenic trioxide/itraconazole in patients with refractory basal cell carcinoma.

SECONDARY OBJECTIVES:

I. To determine if this treatment is associated with a reduction in Gli messenger ribonucleic acid (mRNA) levels in tumor and/or normal skin biopsy samples, when compared to baseline levels.

OUTLINE:

Patients receive arsenic trioxide orally (PO) and itraconazole PO daily for 50 days, followed by maintenance therapy consisting of 2 weeks off treatment and then 2 weeks on treatment for up to 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Basal cell carcinoma (BCC)
* Patients ineligible for curative locoregional treatment and have either progressed on, did not tolerate, unwilling to try or ineligible for investigational smoothened antagonist such as Erivedge or Odomzo
* Life expectancy estimate > 3 months
* Performance status Eastern Cooperative Oncology Group (ECOG) 0 to 2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.9 mg/dL
* Corrected QT (QTC) by 12 lead electrocardiography (EKG) < 450 msecs
* Serum potassium, magnesium and calcium levels which fall within normal limits or levels outside the normal range determined not to be clinically significant by the principal investigator (PI)
* Serum prothrombin time, international normalized ratio (INR) and partial thromboplastin times which fall within normal limits or levels outside the normal range determined not to be clinically significant by the PI
* Ability to understand and the willingness to sign a written informed consent document
* Females and males of reproductive potential must use effective contraception during and after treatment for 6 months

Exclusion Criteria:

* Concurrent use of other investigational agents
* Cardiac arrhythmias
* Receiving potassium wasting diuretics or amphotericin must be noted to have theoretically increased arrhythmia risks with arsenic trioxide (potassium wasting diuretics or amphotericin are not excluded)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, liver disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recurrent seizure history or psychiatric illness/social situations that would limit compliance with treatment requirements
* Currently taking systemic medications that would affect BCC tumors (oral retinoids) or metabolism of itraconazole (anti convulsants and corticosteroids); itraconazole should not be taken with cisapride (Propulsid), dofetilide (Tikosyn), oral midazolam (Versed), nisoldipine (Sular), pimozide (Orap), quinidine (Quinaglute), triazolam (Halcion), or levomethadyl (Orlaam), lovastatin (Mevacor), simvastatin (Zocor), or an ergot medication such as dihydroergotamine (Migranal), ergometrine or ergonovine (Ergotrate Maleate), ergotamine (Ergomar), or methylergometrine or methylergonovine (Methergine)
* History or current evidence of malabsorption or liver disease that would impair the absorption of itraconazole
* History or current evidence of hyperthyroidism that would increase metabolism of itraconazole
* Immunosuppressed patients (cancer, autoimmune disease) or patients taking immunosuppressive drugs
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in Gli levels | Baseline to up to 1 month
  Nonparametric methods (Wilcoxon sign rank test) will be used given then the continuous outcome and small sample size.

SECONDARY OUTCOMES:
Tumor response using Response Evaluation Criteria in Solid Tumors (RECIST) criteria | At 3 months
  Proportion of subjects with complete response, partial response, stable disease, or disease progression by RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, Principal Investigator — Stanford Cancer Institute

IPD SHARING:
Plan to Share IPD: No